CLINICAL TRIAL: NCT04259242
Title: Impact of Scaling and Root Planing on Systemic Inflammation and Serum Bone Resorption Markers in Premenopausal Women With Periodontitis and Low Bone Mineral Density- A Prospective Interventional Study.
Brief Title: SRP, Systemic Inflammation and Serum Bone Resorption Markers Premenopausal Women With Periodontitis and Low BMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pradeep perio
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- premenopausal women with periodontitis (Experimental): Experimental: premenopausal women with periodontitis premenopausal women with chronic periodontitis will be evaluated after SRP for serum bone resorption markers - CTX and inflammatory markers IL-6
  Interventions: Procedure: SRP

INTERVENTIONS:
Procedure: SRP — scaling and root planing with ultrasonic scaler and manual instruments

SUMMARY:
To assess the impact of scaling and root planing on systemic inflammation and serum bone resorption markers in pre-menopausal women with periodontitis

DETAILED DESCRIPTION:
Periodontitis is a chronic multifactorial inflammatory disease associated with dysbiotic plaque biofilms and characterized by progressive destruction of the tooth supporting apparatus. Its primary features include the loss of periodontal tissue support, manifested through clinical attachment loss (CAL) and radiographically assessed alveolar bone loss, presence of periodontal pocketing and gingival bleeding.

Periodontitis is multifactorial inflammatory disease with numerous systemic or local risk factors playing a part in its clinical sequences. Periodontitis causes increased local inflammation as well as contributes to systemic inflammation with an increase in the levels of local and systemic inflammatory mediators including tumor necrosis factor alpha (TNF-α), interleukin-1 and interleukin-6 (IL-6).

Osteoporosis is a systemic skeletal disease characterized by low bone mass and microarchitectural deterioration of bone tissue, with a consequent increase bone fragility and susceptibility to fracture.

The development of osteoporosis occurs through spontaneous increase in pro-inflammatory and pro-osteoclastic cytokines such as , IL-6 and IL-1 β that activates receptor activator of nuclear factor-Kb ligand (RANKL) leading to an enhanced ability of osteoclasts to resorb bone.

The Studies on systemic influence of periodontitis have suggested that locally produced proinflammatory cytokines such as IL-1β , TNF-α and IL-6 may be released into circulation. Most studies shows that IL-6 and TNF-α is major cytokine responsible for resorption of bone in osteoporosis and increase of bone turnover markers. Periodontitis is chronic inflammatory disease characterized by destruction of tooth supporting tissues by virtue of the immunologic response to bacterial challenge originating from dental plaque. In Periodontitis, the increased released of proinflammatory cytokines such as TNF- α, IL-1β, and IL-6 in systemic circulation which causes increase in systemic bone loss through their osteoclastic activity. The systemic inflammation and rate of bone loss is measured by systemic inflammatory and bone resorption markers respectively.

Till date there is no conclusive interventional study done on impact of management of periodontitis on systemic inflammation and bone resorption markers(serum CTX) in pre-menopausal women with periodontitis .

METHODOLOGY The study will be conducted as follows This prospective interventional study will be conducted in the department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences (PGIDS), Rohtak.

Periodontitis patients will be recruited from the outpatient department of PGIDS, Rohtak.

Sample Size calculation:

Sample size was calculated using G power software using t test to compare difference between two matched (dependent) means . Total sample size was calculated as 19. A total of 24 patients will be recruited expecting a 25% dropout rate.

Periodontal parameters:

At baseline, periodontal parameters plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing depth (PD), clinical attachment loss (CAL) will be assessed at six sites (disto-buccal, mid-buccal, mesio-buccal, mesio-lingual, mid-lingual and disto-lingual) per tooth excluding third molars. Periodontal examination would be performed at baseline and 8 weeks after scaling and root planing.

Periodontal therapy:

After recording periodontal parameters at baseline, oral hygiene instructions would be given and scaling and root planning would be done. Patient would be recalled at after 8 weeks of complete scaling and root planing.

Blood collection and serum analysis:

For assessing markers of systemic inflammation and bone resorption, serum samples will be collected from venipuncture in antecubital fossa at 8 hours and after an overnight fasting for all subjects at baseline in individuals meeting the inclusion criteria. Serum samples would again be analyzed for systemic markers at 8 weeks after scaling and root planing in individuals who have bleeding on probing (BOP) less than 10% of the total sites.

Parameters of systemic inflammation that would be assessed:

Interleukin-6 (IL-6) Total leukocyte count(TLC) Differential leukocyte count (DLC) Platelet count Neutrophil/lymphocyte ratio (N/L) mean platelet volume platelet distribution width

Systemic marker of bone resorption that would be analyzed:

Serum C-terminal telopeptide of type 1 collagen (s-CTX-1)

Anthropometric parameter that would be measured:

Body Mass Index (BMI) calculated as weight/height 2 (Kg/m2)

METHOD:

Pre-menopausal women having stage 2 or stage 3 periodontitis would be enrolled to participate in the study. Those who fulfill the inclusion criteria would be enrolled in the study clinical periodontal parameters(CAL,PD,and BOP) would be recorded and venous blood samples for measuring serum levels of IL-6, and serum CTX-1 would be collected. Scaling and root planing would be performed in all cases.

Patients would be re-evaluated after 8 weeks for recording all the periodontal parameters and systemic inflammation (IL-6 ) and systemic resorption marker (serum CTX-1 ).

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women ( Pre-menopause was defined as women above 40 years of age with regular menstruation).
* Periodontitis with 20 or more natural teeth (excluding third molars). Periodontitis criteria
* Periodontal classification stage 2 and stage 3 ( 2017 World Workshop on classification of Periodontal and peri-implant Disease and conditions)
* Bleeding on probing with more than 30% site ( 2017 World Workshop on classification of Periodontal and peri-implant Disease and conditions)

Exclusion criteria:

* Systemic inflammatory diseases known to affect BMD such as rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, and chronic obstructive pulmonary disease.
* History of diabetes, metabolic bone disease, thyroid and parathyroid disease, and gastrointestinal disorders
* Treatment with the following drugs in the previous 3 months : steroids, immunosuppressants, antibiotics, NSAIDs ,statins, lipid lowering drugs, anticonvulsants, thiazide diuretic agents, anti-coagulants, oral contraceptive drugs or any other host modulatory drug
* Recent history or presence of acute or chronic infection
* Previous history of treatment for osteoporosis/osteopenia.
* Current or former smokers or use of smokeless tobacco in any form
* Periodontal treatment within past 1 year prior to inclusion into the study.
* pregnant and lactating mothers.

Ages: 40 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in serum IL-6 . | 8 weeks
  change in serum IL-6
serum CTX-1 | 8 WEEKS
  Change in serum CTX-1

SECONDARY OUTCOMES:
Platelet count | 8 weeks
  Number of platelets
PMV | 8 weeks
  Platelet Mean Volume
PDV | 8 weeks
  Platelet Distribution Width

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Sharma, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol